CLINICAL TRIAL: NCT06738121
Title: Cosmetic Outcomes of Umbilical Hernia Incisions; A Randomized Controlled Trial
Brief Title: Cosmetic Outcomes of Umbilical Hernia Incisions
Acronym: UHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Tolulope Oyetunji, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003347
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Umbilical Hernia
Keywords: Umbilical Hernia
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Infra-umbilical incision (Active Comparator): Patients randomized to this arm with have the traditional curvilinear infra-umbilical incision
  Interventions: Procedure: Infra-umbilical incision
- Vertical Trans-umbilical Incision (Active Comparator): Patients in this arm will have the cranio-caudal vertical incision right through the umbilicus for the repair of the umbilical hernia
  Interventions: Procedure: Transumbilical incision

INTERVENTIONS:
Procedure: Infra-umbilical incision — Traditional curvilinear infra-umbilical incision is used to repair the umbilical hernia
  Arms: Traditional Infra-umbilical incision
Procedure: Transumbilical incision — The incision for the repair of the umbilical hernia will be carried through the umbilicus itself.
  Arms: Vertical Trans-umbilical Incision

SUMMARY:
This will be a single institution, prospective, randomized controlled trial. Patients presenting as an outpatient for repair of umbilical hernias who meet our inclusion criteria, whose parents provide permission to participate in the study, will receive the umbilical hernia repair that they are randomized to. The appropriate data will be collected on day of surgery, and patients will be followed with a delayed parental submission of incisional photograph.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with umbilical hernia that is <1.5cm in size based on physical exam for outpatient repair
* Treated at CMH Adele Hall or CMHK from 09/11/24 - 09/11/25
* Subjects <10 years of age

Exclusion Criteria:

* Umbilical hernia > 1.5 cm in size
* Patients with prior umbilical surgery
* Subjects ≥10 years of age

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Cosmetic Outcome | 4 - 6 weeks and 2 years post operation
  Cosmetic appearance of incision will be measured using the Pediatric Scar Assessment Questionnaire (PSAQ) filled out by patients and a modified version filled out by an independent assessor .

SECONDARY OUTCOMES:
Operative times | Up to 2 years
  This will evaluate operative time for each procedure in minutes
Surgical site infections | 30 days
  Assess the rate of surgical site infections in each arm of the study
Wound complications | 30 days
  Evaluate wound complication including wound breakdown and wound dehiscence
Recurrence | 2 years
  Recurrence of the umbilical hernia will be calculated as a rate in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Tolulope A Oyetunji, MD, MPH, MBA, Principal Investigator — Division Chief, Pediatric General Surgery
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No